CLINICAL TRIAL: NCT06546631
Title: Investigating Mechanistic Predictors of Interpatient Variability and Temozolomide (TMZ) Induced Haematological Toxicity for Glioma Patients
Acronym: Improve TMZ
Status: Recruiting | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: University Hospital Waterford (Other)
Responsible Party: Sponsor
Other Study IDs: 24010
Record Dates: First submitted 2024-07-29; First posted 2024-08-09 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, saliva and blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Temozolamide treatment: Patients who are being started on Temozolamide treatment for high-grade glioma. Patients will provide blood, saliva and stool samples.
- Temozolamide toxicity: Patients who have developed dose-limiting haematological toxicity during treatment with TMZ for a high grade glioma. Patients will provide blood, saliva and stool samples

SUMMARY:
A medication called temozolomide has been used for many years in the treatment of high-grade gliomas, which are tumours that originate in the brain. While this drug is the normal treatment for high-grade glioma, a number of patients develop a side-effect which results in low levels of some important blood cells, such as platelets or white blood cells. If this side-effect occurs, treatment with temozolomide may have to be stopped or paused, which may affect how well this treatment works.

At present, it is unknown why some patients develop this side effect and others do not. It is known that patients with a higher concentration of temozolomide in their blood are at an increased risk of developing this toxicity. There may be some factors associated with the movement of the drug in the body or the removal of the drug from the body which may affect the concentration of temozolomide in blood. There are many factors which may be involved, including genes, other medicines that are taken, how well kidneys and liver are working or even the microbiome (which is the bacteria in the gut).

This study is being done to find out what these factors could be. In the future, this may lead to medical care teams being able to predict which patients are at higher risk of side-effects, allowing them to implement measures to reduce the risk of this occurring.

DETAILED DESCRIPTION:
Concurrent (with radiotherapy) and adjuvant temozolomide (TMZ) is the standard of care treatment for high grade glioma, however, severe haematological toxicity is a major dose limiting factor, impacting 16-45% of patients in different studies. The investigators hypothesize that mechanistic factors such as genetic polymorphisms, renal function or other patient factors such as sex, concomitant medications or the microbiome result in this interpatient variability in toxicity. This study aims to develop a pharmacokinetic model of temozolomide to test the effect of these potential covariates on TMZ concentration (Part A) in patients with brain tumours being treated with TMZ. Using this model, the investigators aim to assess patients who develop haematological toxicity from TMZ for mechanistic predictors of this toxicity (Part B).

The investigators hypothesise that the development of severe TMZ-induced haematological toxicity is due to higher exposure to temozolomide in plasma, driven by mechanistic factors, such as pharmacogenomic variants, the microbiome or demographic factors.

ELIGIBILITY:
Part A

Inclusion Criteria:

1. 18 years of age or over
2. Will receive or are currently receiving concurrent phase treatment with TMZ for high grade glioma (WHO Grade 3 or Grade 4 Astrocytoma, Oligodendroglioma or Glioblastoma).
3. Provision of informed consent to participate.

Exclusion Criteria:

a. Patients who, in opinion of supervising clinician, are clinically too unwell to provide informed consent or for whom additional blood samples, or other research samples, would not be indicated or appropriate.

Part B

Inclusion Criteria:

1. 18 years of age or over
2. Receiving or received treatment with TMZ for high grade glioma (WHO Grade 3 or Grade 4 Astrocytoma, Oligodendroglioma or Glioblastoma).
3. Developed any CTCAE Grade ≥3 Haematological Toxicity associated with Temozolomide, and/or any 1 of:

i. Platelet count <100 x 109/L ii. Neutrophil Count <1.0 x 109/L iii. Haemoglobin value <8.0 g/L iv. Omission of daily TMZ dose for ≥3 consecutive days during concurrent phase due to FBC concerns v. Deferral of subsequently due TMZ cycle by ≥7 days during adjuvant phase; vi. Dose reduction or permanent discontinuation of TMZ for reasons of haematological toxicity (as per treating physician discretion); vii. Use of growth factors, platelets or packed-cell transfusions during the course of TMZ.

d. Provision of informed consent to participate.

Exclusion criteria:

a. Patients who, in opinion of supervising clinician, are clinically too unwell to provide informed consent or for whom additional blood samples, or other research samples, would not be indicated or appropriate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients under the care of a medical oncologist attending a hospital clinic for the treatment of their high grade glioma
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Determine potential predisposing factors for severe haematological toxicity from temozolamide | On study registration
  Analysis of pharmacogenes
Determine potential predisposing factors for severe haematological toxicity from temozolamide | Baseline and study completion, an average of 9 months
  Microbiome analysis of stool bacterial composition

SECONDARY OUTCOMES:
Assess duration of haematological toxicity from temozolamide | Up to 12 months
  Duration measured in time (days/weeks).
Assess severity of haematological toxicity from temozolamide | Up to 12 months
  Severity measured by Common Terminology Criteria for Adverse Events (CTCAE) Grade (grades range from 1-5, with higher grades indicating higher severity).
Assess the impact of haematological toxicity on patients | Up to 12 months
  Number of blood transfusions required as a result of the haematological toxicity
Assess the impact of haematological toxicity on patients | Up to 12 months
  Number of platelet transfusions required as a result of the haematological toxicity
Assess the impact of toxicity on patients distress tool scores | On date of study registration
  The European Organisation for Research and Treatment of Cancer (EoRTC) Quality of Life questionnaires for cancer patients (C-30, scores range from 30-126). Higher scores indicate lower quality of life.
Assess the impact of toxicity on patients quality of life scores | On date of study registration
  The European Organisation for Research and Treatment of Cancer (EoRTC) Quality of Life questionnaires for cancer patients brain-specific module BN-20 (scores range from 20-80). Higher scores indicate lower quality of life.
Assess the impact of toxicity on patients distress tool scores | On date of study registration
  The National Comprehensive Cancer Network distress thermometer (scores range from 0-10). Higher scores indicate more extreme distress.
Overall survival | From date of study registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Hospital, Cork, Ireland